CLINICAL TRIAL: NCT03731793
Title: Efficacy and Safety of Non-animal Chondroitin Sulphate Supplementation in the Treatment of Moderate Knee Osteoarthritis in a Group of Overweight Subjects: a Randomized, Double Blind, Placebo-controlled Study.
Brief Title: Efficacy of Non-animal Chondroitin Sulphate for Overweight Subjects With Knee Ostoarthritis.
Acronym: NACSKO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Collaborators: Gnosis SpA (Unknown)
Responsible Party: Principal Investigator, Mariangela Rondanelli, MD, Associate Professor, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8810/02112017
Record Dates: First submitted 2018-10-31; First posted 2018-11-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Knee Osteoarthritis
Keywords: non-animal chondroitin sulphate; knee osteoarthritis; overweight
MeSH Terms: conditions — Osteoarthritis, Knee; Overweight

STUDY DESIGN:
Intervention Model Description: Double-blind randomized placebo controlled study. 90 days of treatment with 600 mg/d of non-animal Chondroitin Sulphate or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Full randomization and full blind study. Intervention was named by "integratore A" and "integratore B"
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): Placebo. For 90 days one capsule/day.
  Interventions: Other: Placebo
- Intervention Group (Experimental): 600 mg/day of non-animal Chondroitin Sulphate. One capsule/day for 90 days.
  Interventions: Biological: Non-Animal Chondroitin Sulphate

INTERVENTIONS:
Biological: Non-Animal Chondroitin Sulphate — Mythocondro® is an ichthyic-like chondroitin sulfate produced by chemical sulfation of a non-sulfated chondroitin backbone obtained by thermo-acid hydrolysis of the capsular polysaccharide naturally produced by an Escherichia coli strain.
  Arms: Intervention Group
Other: Placebo — Placebo
  Arms: Placebo Group

SUMMARY:
Knee osteoarthritis (OA) is predicted to become the fourth leading cause of disability worldwide by 2020. and is estimated to affect more than 40 million people in Europe and 4 million people in Italy. OA has multifactorial etiology and obesity is one of the most important risk factor for knee Regarding therapy of OA in 2014, the European Society for Clinical and Economic Aspects of Osteoporosis and Osteoarthritis (ESCEO) published a treatment algorithm for the management of knee OA. In Step 1 of the treatment, it is recommended to initiate therapy with chronic symptomatic slow-acting drugs for osteoarthritis (SYSADOAs). Among SYSADOAs, the evidence is greatest for the effect of chondroitin sulfate (CS).

Sixty overweight subjects with knee osteoarthritis (OA) were recruited and randomly allocated to a group of treatment with 600 mg/d of non-animal Chondroitin sulphate (CS) or to a placebo group.

These measurements were considered:

Tegner Lysholm Knee Scoring (TLKS), Western Ontario and McMaster Universities Arthritis (WOMAC) index and Visual Analogue Scale (VAS) for pain were analyzed at time 0 and at 4 and 12 weeks. Health-related quality of life by ShortForm36, inflammation by C-Reactive Protein (CRP) and Erythrocyte Sedimentation Rate (ESR) were also evaluated, together with a body composition assessment performed by DXA.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian subjects, males and females, with the following characteristics were included in the trial and randomly assigned to the experimental group (N=30) or a control group (N=30): Individuals overweight (BMI > 25 kg/m2), aged 40-74.; Mobility impairment, joint discomfort or established moderate knee OA (classification 1-3 according to Kellgren and Lawrence system for classification of knee OA).

Exclusion Criteria:

* Anyone with evidence of heart disease, kidney or liver disease, or any other disease that might influence the results of the study was excluded.

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-10-20 (Actual)

PRIMARY OUTCOMES:
Change in Generic Pain (VAS) | 0, 30, 90 days
  Pain intensity measured both at motion and at rest, using the Visual Analogue Scale (VAS). VAS measures a characteristic or attitude ranging across a continuum of values and cannot be directly measured. For example, the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks. The results are showed with a scale 0-10. 0 means no pain and 10 high pain. A VAS reduction is expected only in treatment group.
Change in Knee Pain (WOMAC) | 0, 30, 90 days
  Assessment of knee pain by WOMAC (Western Ontario and McMaster Universities Arthritis) Index. The WOMAC pain scale consists of five questions that assess pain while walking on a flat surface, going up or down stairs, in bed at night, sitting or lying, and standing upright. The responses are recorded on a five-point Likert scale, with a higher score representing a greater level of pain. This scale is valid and reliable in hip and knee OA populations. A significant decrease in expected in treatment group.
Change in Knee Functionality (TLKS) | 0, 30, 90 days
  Tegner Lysholm Knee function Scoring (TLKS). Each patient completed a self-report questionnaire, TLKS, related to knee symptoms and function. It includes eight items: Limp, Support, Locking, Instability, Pain, Swelling, Stair climbing and Squatting. Each possible response to the items gives an arbitrary score on an increasing scale with a maximum of 100, a higher score representing a higher ability. An increase in expected in treatment group.

SECONDARY OUTCOMES:
Change in Quality of Life (SF-36) | 0, 30, 90 days
  Health-related quality of life, recorded by the Short Form 36 Health questionnaire (SF-36), a generic measure of health status designed for use in population surveys which consider body pain as a dimension of health status. This is a self-reporting questionnaire and outcomes are measured with 8 numbers that express 8 different aspects of quality of life. Scoring 36-Item Health Survey is a two-step process. First, precoded numeric values are recoded per the given scoring key. all items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. In step 2, items in the same scale are averaged together to create the 8 scale scores. Hence, scale scores represent the average for all items in the scale that the respondent answered.
Change in Inflammatory Markers circulating levels (CRP, ESR) | 0, 30, 90 days
  Inflammation markers in plasma: C-reactive protein (CRP), erythrocyte sedimentation rate (ESR). High-Sensitivity CRP was determined by immunonephelometry while the erythrocyte sedimentation rate (ESR) was analyzed by capillary photometry.
Change in total Fat Mass, Total Free Fat Mass and Visceral adipose tissue (DXA) | 0, 30, 90 days
  Body composition by dual-energy X-ray absorptiometry (DXA). Body composition was measured at baseline by DXA, using a Lunar Prodigy DEXA (GE Medical Systems, Waukesha, WI). Free Fat mass, Fat mass and visceral fat data were derived from DXA using the DXA Prodigy enCORE software (version 17; GE Healthcare).

CONTACTS AND LOCATIONS:
Overall Officials: Mariangela Rondanelli, Professor, Study Director — IRCCS Mondino Foundation, Pavia
Locations (1):
- Geriatric physical medicine and rehabilitation division at the Istituto Santa Margherita - Azienda di Servizi alla Persona di Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No
Data are planned to be available for Gnosis SpA and together with the study pubblication. IPD will be not available for other researchers.